CLINICAL TRIAL: NCT03885492
Title: The Baby-Saver Kit: Development and Evaluation of a Novel Device for Affordable Neonatal Resuscitation in a Low-income Region in Africa
Brief Title: The Baby-Saver Kit: Clinical Testing of a Device for Neonatal Resuscitation With Intact Cord in Uganda
Acronym: BabySaver
Status: Terminated | Type: Observational
Why Stopped: This was part of a University of Liverpool PhD programme, but PI suspended by University and left the programme. Also dismissed by sponsoring organisation SAfRI. Likely unreliable data so project abandoned with no plans to publish.
Sponsor: Sanyu Africa Research Institute (Other)
Collaborators: University of Liverpool (Other); Grand Challenges Canada (Other); Mbale Regional Referral Hospital (Other); Makerere University (Other)
Responsible Party: Sponsor
Other Study IDs: BabySaver-01
Record Dates: First submitted 2019-03-16; First posted 2019-03-21 (Actual); Last update posted 2023-10-25 (Actual); Status verified 2023-10

CONDITIONS: Birth Asphyxia; Neonatal Resuscitation; Maternal Distress
MeSH Terms: conditions — Asphyxia Neonatorum

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
To examine the usability, safety and acceptability of the BabySaver kit: a novel device for neonatal resuscitation in a low-income region in Africa

DETAILED DESCRIPTION:
The BabySaver kit will be used for any delivery in which the baby requires resuscitation according to the hospital policy, national guidelines(Ministry of Health, 2016) and WHO policy(World Health Organization, 2014)

The target sample size for observation will be 30 babies requiring resuscitation at Mbale Regional Referral Hospital Delivery suite.

The researchers will observe midwives and mothers during the process of resuscitation. This will be a non-participant observation. The researchers will collect data on: demographics, the timing of cord clamping, time to establish ventilation, intervention provided on the kit, post-resuscitation temperature, need to move the baby to provide extra care, and notes of the ease of use or challenges experienced with the kit. The researchers will ask health workers for their views of the usability of the kit in comparison to the equipment in current use.

The researchers have developed a usability checklist to assess how health workers are using the BabySaver kit.

ELIGIBILITY:
Inclusion Criteria:

* As this is the first delivery suite to use the kit in a clinical setting, we will include only low-risk babies in this study. Every low-risk birth that will need neonatal resuscitation will be selected and observations made for the use of the BabySaver resuscitation kit.

Exclusion Criteria:

* High risk deliveries will be excluded, namely

  * babies born before 34 weeks' gestation,
  * babies with life threatening malformations or significant intrapartum asphyxia

Ages: 15 Years to 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: The BabySaver kit will be used for any delivery in which the baby requires resuscitation according to the hospital policy, national guidelines(Ministry of Health, 2016) and WHO policy(World Health Organization, 2014). These include
  * Deliveries before 37 weeks of gestation
  * Deliveries with evidence of fetal distress from fetal monitoring
  * Instrumental deliveries
  * Deliveries in which there is a possibility of a life-threatening malformation
  * Deliveries in which meconium stained liquor has been noted.
Sampling Method: Non-Probability Sample
Enrollment: 47 (Actual)
Dates: Start 2020-11-01 (Actual); Primary Completion 2021-04-01 (Actual); Study Completion 2021-04-01 (Actual)

PRIMARY OUTCOMES:
Change from 10 minutes in post-resuscitation temperature at 30 minutes | Between 10 and 30 minutes after birth
  The researcher will measure post resuscitation temperatures at 10, 20 and 30 minutes afterbirth for babies not admitted to the neonatal unit after using the BabySaver.
Number of procedures performed to newborns while on the BabySaver kit | at birth, upto 30 minutes
  The researcher will list any resuscitation procedures or interventions provided to the newborns on the kit.
change from childbirth in post-resuscitation temperature at admission to Neonatal unit. | Upon admission to Neonatal unit, up to 1 hour after birth
  For babies admitted to the neonatal unit, the baby's temperature will be measured on admission to the Neonatal unit

SECONDARY OUTCOMES:
change from birth in Apgar score at 5 minutes | upto 5 minutes
  Apgar score will be recorded at 1 minute and 5 minutes. Resuscitation of babies at birth will be performed in line with existing hospital guidelines.
Demographic assessments | baseline
  Researchers will collect both mother's (age, marital status, education, occupation) and baby's demographic characteristics (sex, birth weight, gestation at birth).
Design assessments transcripts | uptown 2 months
  Researchers will collect data about design and practical aspects of the BabySaver kit from mothers, carers, midwives and doctors in form of audio and video recordings and extra notes. These will be transcribed verbatim for analysis using an NVivo qualitative software.

CONTACTS AND LOCATIONS:
Overall Officials: Andrew D Weeks, MD, Study Chair — University of Liverpool
Locations (1):
- Mbale Regional Referral hospital, Mbale, Uganda